CLINICAL TRIAL: NCT00001405
Title: Recruitment and Apheresis Collection of Peripheral Blood Hematopoietic Stem Cells, Mononuclear Cells and Granulocytes
Status: Recruiting | Type: Observational
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Other Study IDs: 940073; 94-I-0073
Record Dates: First submitted 1999-11-03; First posted 1999-11-04 (Estimated); Last update posted 2026-01-05 (Actual); Status verified 2025-08-28

CONDITIONS: Granuloma; Granulomatous Disease, Chronic; Leukocyte Disease; Genetic Disease, X-Linked; Genetic Disease, Inborn
Keywords: Chronic Granulomatous Disease; CD34 Cells; Infection; Nadph Oxidase; Healthy Volunteer; Natural History; Normal Volunteer
MeSH Terms: conditions — Granuloma; Granulomatous Disease, Chronic; Genetic Diseases, X-Linked; Genetic Diseases, Inborn; Infections

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Healthy Volunteers: Healthy Adult Volunteers
- Patients: Pts with PID or other blood disorder or clinical history consistent with PID or other blood disorder. Pts are able to volunteer as patient for research collection only per PI discretion.

SUMMARY:
The research goal of this study is to obtain CD34+ hematopoietic stem cells (HSC) from peripheral blood and/or bone marrow, and Mononuclear Cells (lymphocytes and monocytes), and granulocytes (grans) from peripheral blood that will be used in the laboratory and/or in the clinic to develop new cell therapies for patients with inherited or acquired disorders of immunity or blood cells. Development of novel cellular therapies requires access to HSC, Mononuclear Cells and/or granulocytes as the essential starting materials for the pre-clinical laboratory development of gene therapies and other engineered cell products. HSC or blood cells from healthy adult volunteers serve both as necessary experimental controls and also as surrogates for patient cells for clinical scale-up development. HSC or blood cells from patients serve both as the necessary experimental substrate for novel gene therapy and cellular engineering development for specific disorders and as pre-clinical scale up of cellular therapies. Collection of cells from adult patients collected in the NIH Department of Transfusion Medicine (DTM) under conditions conforming to accepted blood banking clinical practice may also be used directly in or cryopreserved for future use in other NIH protocols that have all required regulatory approvals allowing such use. In summary, the research goal of this protocol is the collection of HSC or blood cells that may be used for both laboratory research and/or for clinical treatment in other approved protocols.

DETAILED DESCRIPTION:
The research goal of this study is to obtain CD34+ hematopoietic stem cells (HSC) from peripheral blood and/or bone marrow, and Mononuclear Cells (lymphocytes and monocytes), and granulocytes (grans) from peripheral blood that will be used in the laboratory and/or in the clinic to develop new cell therapies for patients with inherited or acquired disorders of immunity or blood cells. Development of novel cellular therapies requires access to HSC, Mononuclear Cells and/or granulocytes as the essential starting materials for the pre-clinical laboratory development of gene therapies and other engineered cell products. HSC or blood cells from healthy adult volunteers serve both as necessary experimental controls and also as surrogates for patient cells for clinical scale-up development. HSC or blood cells from patients serve both as the necessary experimental substrate for novel gene therapy and cellular engineering development for specific disorders and as pre-clinical scale up of cellular therapies. Collection of cells from adult patients collected in the NIH Department of Transfusion Medicine (DTM) under conditions conforming to accepted blood banking clinical practice may also be used directly in or cryopreserved for future use in other NIH protocols that have all required regulatory approvals allowing such use. In summary, the research goal of this protocol is -the collection of HSC or blood cells that may be used for both laboratory research and/or for clinical treatment in other approved protocols.

Participants include: 1. Adult patients with any primary immune deficiency (PID) or other blood disorder where collection is both for clinical use in another approved treatment protocol to benefit the patient and for laboratory research; 2. Adult patients with any primary immune deficiency (PID) or blood disorder where collection is for laboratory research use only. 3. Healthy adult volunteers where the collection is for laboratory research use only.

The majority of subjects will have HSC collected from peripheral blood by apheresis. Daily subcutaneous injections of G-CSF (granulocyte colony stimulating factor/filgrastim) for 5 to 6 days is a standard of care method used to mobilize HSC to the peripheral blood prior to apheresis, and will be used for most subjects. Plerixafor (Mozobil) is approved as standard of care for use in combination with G-CSF to mobilize HSC.

Some adult patients will have a clinical scale aspiration collection of bone marrow to obtain HSC for clinical use in another approved treatment protocol. Some adult participants may have a small sample needle aspiration collection of bone marrow obtained for laboratory research purposes only.

Mononuclear cells and/or Granulocytes (gran) will be collected from peripheral blood by apheresis following no stimulation, using G-CSF alone, or a using a combined single dose of G-CSF (480mcg) and Dexamethasone (8mg) prior to collection as is the standard of care pre-treatment used in the NIH DTM for collection of granulocyte transfusions from healthy donors.

As noted, HSC, mononuclear cells, and gran collection from patients with PID or other blood disorders may be used for laboratory research or may be designated for future clinical treatment of the patient under separate treatment protocol. HSC, mononuclear cells, and gran collection from healthy volunteers will be designated entirely for laboratory research.

HSC will be used for the following clinical purposes, where clinical treatments would occur under separate IRB approved protocols: 1. Autologous HSC from patients may be genetically modified and infused into the patient for treatment of an infection or the underlying disease (Gene therapy); 2. Autologous HSC from patients may serve as back up (rescue product) for patients undergoing matched unrelated donor transplantation or haploidential related or unrelated donor transplantation.

Mononuclear Cells (lymphocytes and monocytes) and granulocytes will be used for the following clinical purposes, 1. Autologous lymphocytes may be genetically modified and infused into the patient for treatment of an infection or the underlying disease (Gene therapy); 2. Autologous lymphocytes, monocytes and granulocytes (neutrophils) may be transfected with mRNAs to transiently express a therapeutic protein for treatment of an infection or the underlying disease (Gene therapy).

HSC, lymphocytes, monocytes and granulocytes will be used for laboratory research studies that include: Delineating the pathophysiology of inherited immune deficiencies; Delineating the physiology of and improving engraftment of hematopoietic stem cells; Determining how hematopoietic stem cells may be maintained in ex vivo culture without losing pluripotent potential; Delineating the molecular mechanisms responsible for lineage specific differentiation; Developing efficient methods for gene transfer into hematopoietic stem cells for corrective gene therapy; Developing methods for restoration of function in defective peripheral blood monocytes and/or granulocytes; Further characterization of peripheral blood monocytes and/or granulocytes from patients with PID.

ELIGIBILITY:
* ELIGIBILITY CRITERIA:

Patients (Patients with a genetically defined PID or other blood disorder or clinical history consistent with PID or other blood disorder)

1. Patients will have a genetically defined PID or have a clinical history of recurrent infections or other problems suggestive of PID or other blood disorder, must be 18-70 years of age,
2. Some patients may have active bacterial or fungal infection at the time of study entry.
3. Preserved renal function (creatinine less than or equal to 2.5 mg/dL; less than or equal to 3+ proteinuria); preserved hepatic function (bilirubin less than or equal to 2.0 mg/dl); preserved hematologic function (WBC greater than or equal to1000/mm^3;granulocytes greater than or equal to 500/mm^3; platelets greater than or equal to 100,000; hematocrit greater than or equal to 25). Of note, patients with PID often have associated chronic thrombocytopenia. Patients with stable chronic thrombocytopenia will be eligible for collection, at the investigator s discretion, with the caveat that patients with platelet count <40,000 the day prior to collection will be transfused with platelets on the morning of collection. Platelets may also be given to these patients following the collection if medically indicated..
4. Patients of childbearing potential may be entered if using effective contraception and having a negative serum or urine pregnancy test within one week of beginning G-CSF administration.
5. Patients may remain on their regimen of prophylactic treatments as deemed necessary by the investigator.
6. Willingness to allow blood cell samples to be stored
7. Willingness to allow blood and/or bone marrow samples to be modified to iPS cells

Healthy Adult Volunteers

1. Healthy adults aged 18-65 without active current infection or history of recurrent infection,
2. Weighs at least 50kg.
3. Normal renal function (creatinine less than or equal to 1.5 mg/dL; less than or equal to 1+ proteinuria); normal hepatic function (bilirubin less than or equal to 1.5 mg/dL); normal hematologic function (WBC greater than or equal to 2500/mm^3; granulocytes greater than or equal to 1200/mm^3; platelets greater than or equal to 120,000; hematocrit greater than or equal to 38).
4. Normal female volunteers of childbearing potential may be entered if using effective contraception and having a negative serum or urine pregnancy test within one week of beginning GCSF administration.
5. Willingness to allow blood cell samples to be stored
6. Willingness to allow blood and/or bone marrow samples to be modified to iPS cells

For PBMCs and grans collections, adult subjects with known genetic mutations may participate as healthy volunteers for research purposes as long as the other criteria listed above are fulfilled.

EXCLUSIONS:

Patients

1. Patients who are hemodynamically unstable (systolic or diastolic blood pressure fall of 20 mm Hg from the stable patient s baseline measurement) or requiring mechanical respiratory assistance are excluded.
2. Female patients who are pregnant or lactating as determined by history and/or positive pregnancy test are excluded.
3. Must be negative by routine blood donor eligibility testing criteria including tests for syphilis (RPR) and TTV Donor Transplant Panel testing (list is modified periodically, but may include hepatitis B and C, HIV and HTLV, T. cruzi). This does not apply to leukapheresis patients, as these tests are not required by DTM.

   1. XSCID patients do not make antibodies and false positives may occur because they receive periodic infusions of pooled donations of IVIG. We have observed positive anti-HBc testing in these patients. If this occurs, more specific DNA or antigen testing will be done and must be negative.
   2. Patients with CGD and other patients with autoimmunity as part of their PID phenotype may have false positive antibody tests and if this occurs more specific DNA or antigen testing will be done and must be negative.
   3. Autologous HSC Transplant patients - may be positive for Hepatitis B and C if the investigator deems it necessary to be collected and used as a safety back-up

Healthy Volunteers

1. Active bacterial, fungal or viral infection as evidenced by history, physical exam (temperature >38 degress C), or WBC >9000 are excluded.
2. Females who are pregnant or lactating as determined by history and/or pregnancy test are excluded.
3. Must be negative by routine blood donor eligibility testing criteria, including tests for syphilis (RPR) and TTV Recipient Transplant Panel (list is modified periodically, but may include hepatitis B and C, HIV and HTLV, T. cruzi) This does not apply to leukaphersis patients, as these tests are not required by DTM policy.
4. Someone without peripheral venous access in arm veins adequate for apheresis (healthy volunteers only).
5. If in the opinion of the investigator participation in this study places the healthy adult volunteer at undue risk.

Patients being considered for clinical scale bone marrow harvesting

1. Who are unable to lie prone during the bone marrow harvesting procedure.
2. Who are unable to tolerate general anesthesia during the bone marrow harvesting procedure.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients with PID or other blood disorders Healthy adult individuals volunteering for research donation
Sampling Method: Non-Probability Sample
Enrollment: 850 (Estimated)
Dates: Start 1994-02-27 (Actual)

PRIMARY OUTCOMES:
Mobilize to peripheral blood and apheresis collect CD34+PBSC of PID patients for clinical treatment and in part (or entirely) for laboratory research | 1/1/2025
  1. To efficiently and safely mobilize to the peripheral blood and apheresis collect CD34+ PBSC patients with any inherited primary immune deficiency (PID) or other blood disorders where PBSC from these patients may be designated entirely or in part for future clinical treatment of the patient
Mobilize to the peripheral blood and apheresis collect CD34+PBSC from healthy volunteers for research | 1/1/2025
  2. To efficiently and safely mobilize to the peripheral blood and apheresis collect CD34+ PBSC from healthy volunteers, which will be designated entirely for laboratory research.
Mobilize to peripheral blood mononuclear cells and granulocytes | 1/1/2025
  3.To efficiently and safely collect peripheral blood mononuclear cells and granulocytes from adult subjects with chronic granulomatous disease or other PID affecting granulocyte function, or from adult healthy donors volunteers for preclinical cell therapy studies, following either no stimulation, G-CSF or dexamethasone alone, or combined single dose G-CSF and dexamethasone as per DTM protocol depending on the number of cells desired.
bone marrow harvest | 1/1/2025
  4.To perform a bone marrow harvest by needle aspiration using standard of medical care methods from adult patients with PID or other blood disorder in sufficient quantity cryopreserved in CC DTM to serve as the source of autologous HSC for gene transfer ex vivo transduction if that patient is enrolled in a separate IRB approved protocol of gene transfer treatment designed to treat the genetically defined type of PID affecting that patient; and the patient has been unable to mobilize and have collected sufficient PBSC to qualify for treatment in that protocol.
bone marrow by needle aspiration | 1/1/2025
  5.To obtain from adult patients with PID or other blood disorder and from adult healthy volunteers a small sample of bone marrow by needle aspiration from bone marrow aspirates, where the purpose for this aspirate is to obtain bone marrow HSC for laboratory research comparing these cells to the biological properties of PBSC.
laboratory studies of PBSC and bone marrow HSC | 1/1/2025
  6.To conduct laboratory studies of PBSC and bone marrow HSC obtained from patients with PID or healthy volunteers in order to: study the functional properties of immune cells arising from hematopoietic stem cells in ex vivo culture systems and in NOD/SCID or NOG mice capable of supporting a human hematopoietic stem cellchimeric marrow xenograft.
laboratory studies of mononuclear cells and granulocytes obtained from patients with PID or healthy volunteers | 1/1/2025
  7.To conduct laboratory studies of mononuclear cells and granulocytes obtained from patients with PID or healthy volunteers in order to: Develop effective methods to restore immunologic function to defective granulocytes/mononuclear cells utilizing mRNA electroporation. Develop methodology of using autologous corrected granulocytes/mononuclear cells for the treatment of infections in immunedeficient patients.

CONTACTS AND LOCATIONS:
Overall Officials: Harry L Malech, M.D., Principal Investigator — National Institute of Allergy and Infectious Diseases (NIAID)
Locations (1):
- National Institutes of Health Clinical Center, Bethesda, Maryland, United States

REFERENCES:
- [Background] Sekhsaria S, Fleisher TA, Vowells S, Brown M, Miller J, Gordon I, Blaese RM, Dunbar CE, Leitman S, Malech HL. Granulocyte colony-stimulating factor recruitment of CD34+ progenitors to peripheral blood: impaired mobilization in chronic granulomatous disease and adenosine deaminase--deficient severe combined immunodeficiency disease patients. Blood. 1996 Aug 1;88(3):1104-12. PMID 8704221
- [Background] Li F, Linton GF, Sekhsaria S, Whiting-Theobald N, Katkin JP, Gallin JI, Malech HL. CD34+ peripheral blood progenitors as a target for genetic correction of the two flavocytochrome b558 defective forms of chronic granulomatous disease. Blood. 1994 Jul 1;84(1):53-8. PMID 7517218
- [Background] Malech HL, Maples PB, Whiting-Theobald N, Linton GF, Sekhsaria S, Vowells SJ, Li F, Miller JA, DeCarlo E, Holland SM, Leitman SF, Carter CS, Butz RE, Read EJ, Fleisher TA, Schneiderman RD, Van Epps DE, Spratt SK, Maack CA, Rokovich JA, Cohen LK, Gallin JI. Prolonged production of NADPH oxidase-corrected granulocytes after gene therapy of chronic granulomatous disease. Proc Natl Acad Sci U S A. 1997 Oct 28;94(22):12133-8. doi: 10.1073/pnas.94.22.12133. PMID 9342375
- See also: NIH Clinical Center Detailed Web Page — https://clinicalstudies.info.nih.gov/cgi/detail.cgi?A_1994-I-0073.html